CLINICAL TRIAL: NCT04697771
Title: The Effect of Telerahabilitation on Fine Motor Skills and Writing Performance in Children With Attention Deficit and Hyperactivity Disorder: A Randomized Controlled Study
Brief Title: Effect of Telerehabilitation on Handwriting Performance in Children With ADHD: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Busra Kaplan Kilic, Occupational Therapist, MSc, Hacettepe University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: E1-20-1038
Record Dates: First submitted 2020-12-28; First posted 2021-01-06 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Handwriting; Telerehabilitation; Fine Motor Skills
Keywords: ADHD; Handwriting; Occupational Therapy; Telerehabilitation
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: Participants will be randomly divided into two groups. The same intervention will be applied to the second group after the first group has received intervention for 8 weeks.
Who Masked: Outcomes Assessor
Masking Description: The person making the first and last outcome assessor does not know which group the participants are from.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): First Evaluation - Fine Motor Skills Training - 8 week - 3 session per week - 40 minute per session - Second Evaluation
  Interventions: Other: Fine Motor Skills Training
- Control Group (No Intervention): First Evaluation - 8 week waiting period - Second Evaluation

INTERVENTIONS:
Other: Fine Motor Skills Training — The fine motor skills training program was planned for the areas of difficulty that children with ADHD experience in the fine motor area as stated in the literature (Lavasani & Stagnitti, 2011). The fine motor goals were organized for 8 weeks, each week including a different fine motor area and practicing handwriting. For each fine motor goal, 3 different activities were identified that did not require materials or could be practiced with materials that could be easily found in each child's home. For example, for the fine motor strengthening goal, three different activities were planned for the same purpose with tools such as play dough, nails, and staples (Case-Smith & O'Brien, 2013). The activities determined each week were repeated three days a week in the same way and applied to all children. Within the 40-minute session, each activity was performed for 10 minutes under the guidance of an expert occupational therapist.
  Arms: Intervention Group

SUMMARY:
This is a randomized controlled study examining the effect of telerehabilitation on fine motor performance and handwriting difficulties experienced by children with attention deficit hyperactivity disorder.

DETAILED DESCRIPTION:
It is planned that 40 children between the ages of 6-8 diagnosed with attention deficit and hyperactivity disorder and their families will participate voluntarily. An informed consent form, BOT-2 and Minnesota Handwriting Test will be sent to volunteer participants via e-mail. An evaluation session on Zoom application will be held for each participant with the participation of the occupational therapist, child and family. After the evaluation, the participants will be randomized and allocated to study and control groups.

Fine motor skills training will be given to the study group 3 sessions a week. The training will be given on the Zoom application and the duration is 8 weeks. At the end of 8 weeks, the evaluation will be done again with BOT-2 and Minnesota Handwriting Test.

The control group will be evaluated with BOT-2 and Minnesota Handwriting Test for the second time after waiting 8 weeks and will receive fine motor skills training.

ELIGIBILITY:
Inclusion Criteria:

* To be in the age range of 6-8,
* Diagnosed with Attention Deficit Hyperactivity Disorder-Predominantly Inattentive subtype according to DSM-5 and ADHD Rating Scale-5,
* Continuing individual education,
* After being informed about the study have agreed to participate in the study.

Exclusion Criteria:

* Children with an additional physical and neurological problem to accompany

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-12-28 (Actual)

PRIMARY OUTCOMES:
Minnesota Handwriting Test | 5 minute
  It evaluates six categories, including legibility, form, alignment, size, spacing, and rate

SECONDARY OUTCOMES:
Bruininks-Oseretsky Motor Proficiency Test- 2 Short Form (BOT-2) | 15 minute
  The test has been produced as a motor function assessment tool that can be applied to children in a short time.
  Fine motor accuracy, fine motor integration, dexterity, bilateral coordination and upper extremity coordination sub-parameters of the test will be applied.

CONTACTS AND LOCATIONS:
Overall Officials: Gonca Bumin, Prof, Study Director — Hacettepe University; Hakan Öğütlü, Msc, Study Director — Ankara City Hospital Bilkent
Locations (1):
- Hacettepe University, Ankara, Ankara - Altındağ, Turkey (Türkiye)

DOCUMENTS (1):
  • Informed Consent Form (2020-09-02): https://cdn.clinicaltrials.gov/large-docs/71/NCT04697771/ICF_000.pdf